CLINICAL TRIAL: NCT04633408
Title: Cultural Adaptation of a Behavioral Intervention for Latino Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Magaly Ramirez, Assistant Professor, School of Public Health, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009534
Record Dates: First submitted 2020-10-30; First posted 2020-11-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Latino; Caregiver; Cultural adaptation
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: A qualitative study, a participatory design study and a randomized pilot study to assess acceptability of an intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The investigators will recruit 15 Latino caregivers for each study arm (total sample size of 30). The sample size was based on a rule of thumb of 12 to 15 participants per group for pilot studies. This group will have access to the app.
  Interventions: Behavioral: STAR-C Virtual Training and Follow-up (STAR-VTF)
- Control (No Intervention): 12 to 15 participants, will not have access to the app.

INTERVENTIONS:
Behavioral: STAR-C Virtual Training and Follow-up (STAR-VTF) — STAR-C Virtual Training and Follow-up (STAR-VTF) is adapted from an evidence-based, in-person program that trains family caregivers to manage BPSD (behavioral and psychological symptoms of dementia)
  Arms: Intervention

SUMMARY:
The overall objectives of the proposed research are to: (i) develop a prototype of a smartphone application (app) that can deliver culturally adapted STAR-C training to Latino caregivers, and (ii) understand the extent to which a STAR-C app is acceptable and potentially effective among Latino caregivers. Achieving these objectives will lay the groundwork for a future full-scale trial to test the STAR-C app with Latino caregivers.

This study aims to: Adapt the STAR-C training to increase cultural relevance for Latino caregivers. The adaptations will focus on incorporating cultural examples, identities, values, beliefs, and practices within the training, as well as using cultural idioms, metaphors, and sayings to compliment explanations. Develop a prototype of a STAR-C app for Latino caregivers. The prototype will be iteratively developed with active participation from Latino caregivers. The final prototype will consist of a fully interactive app that delivers culturally relevant STAR-C training in an engaging and easy to use format. Assess the acceptability and potential effectiveness of the STAR-C app for Latino caregivers. Measures of acceptability will include app usage and perceived ease-of-use and usefulness of the STAR-C app. Measures of potential effectiveness will include changes in caregiver burden and depression.

DETAILED DESCRIPTION:
For aim 1, the investigators plan to recruit 25-30 participants with representation from both caregivers and providers. The investigators will recruit Latino Family Caregivers of persons with ADRD (Alzheimer's Disease and related Dementias). The investigators will recruit providers who work in an organization serving Latino elderly. Participants will be >18 years old.

For aim 2, the investigators will recruit 5 caregivers per session. With three iterative design sessions, the investigators anticipate 15 caregivers in total. The investigators will use the same eligibility criteria described for aim 1.

For aim 3, the investigators will recruit 15 Latino caregivers for each study arm (total sample size of 30). The investigators based the sample size on a rule of thumb of 12 to 15 participants per group for pilot studies. The investigators will use the same eligibility criteria and recruitment strategy described for aim 1

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Family member or close friend of a person with ADRD
* Provide at least eight hours of care per week Speak English or Spanish
* Self-identify as Latino.

Exclusion Criteria:

* Caregiver who has a diagnosis of ADRD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | 2 months
  To assess acceptability, the investigators will measure: (1) app usage. The investigators will obtain data automatically collected by the platform to measure whether caregivers complete the training sessions, how many times caregivers visited the app, and the amount of time between app visits.
Acceptability | 2 months
  To assess acceptability, the investigators will measure (2) perceived ease-of-use. For perceived ease-of-use, the investigators will administer the System Usability Scale. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree (score 5) to Strongly disagree (score 1).
Acceptability | 2 months
  To assess acceptability, the investigators will measure (3) perceived usefulness. For perceived usefulness, the investigators will administer the Perceived Usefulness Scale. It consists of a 6 item questionnaire, all items are measured on a 7-point Likert-type scale ranging from "strongly disagree" (score 1) to "strongly agree" (score 7).
Potential Effectiveness | 2 months
  To assess potential effectiveness, the investigators will measure (1) caregiver burden. For caregiver burden, the investigators will administer the Screen for Caregiver Burden (SCB). The 25-item SCB, provides scores for objective burden (OB; number of potentially negative experiences) and subjective burden (SB; appraised distress in response to the experiences).
  OB scores caregiver experiences that have occurred, regardless of their distress; it scores each item as 0 (did not occur) or 1 (indicating occurrence).
  SB scores evaluate the distress associated with the experiences; it uses five anchor points: 0 = no occurrence of the experience: 1 = occurrence of the experience, but no distress; 2 = occurrence with mild distress; 3 = occurrence with moderate distress; and 4 = occurrence with severe distress.
Potential Effectiveness | 2 months
  To assess potential effectiveness, the investigators will measure (2) caregiver depression. For caregiver depression, the investigators will use the full Patient Health Questionnaire (PHQ)-9. PHQ-9 is the major depressive disorder (MDD) module of the full PHQ. Used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings.
  Scores each of the 9 Diagnostic and Statistical Manual Diploma in Social Medicine (DSM) criteria of MDD as "0" (not at all) to "3" (nearly every day), providing a 0-27 severity score.
  Higher PHQ-9 scores are associated with decreased functional status and increased symptom-related difficulties, sick days, and healthcare utilization.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Alzheimer's Association, Washington State Chapter, Lynnwood, Washington
  - UW Memory and Brain Wellness Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No